CLINICAL TRIAL: NCT00807911
Title: Randomized Phase II Study of Adjuvant Chemotherapy With 5-FU/Leucovorin vs. Oxaliplatin/5-FU/Leucovorin After Preoperative Chemoradiotherapy With Fluoropyrimidines Followed by Surgery in Patients With Locally Advanced Rectal Cancer
Brief Title: Adjuvant Chemotherapy After Preoperative Chemoradiotherapy to Treat Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-0256
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; adjuvant chemotherapy; FOLFOX
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant FL (Active Comparator): FL (5-FU 380 mg/m2, leucovorin 20 mg/m2 on D1-5 q 4 weeks X 4 cycles)
  Interventions: Drug: Adjuvant FL
- Adjuvant FOLFOX (Experimental): FOLFOX (oxaliplatin 85 mg/m2, leucovorin 200 mg/m2 on D1, 5-FU bolus 400 mg/m2 on D1, 5-FU infusion 2400 mg/m2 for 46 hours q 2 weeks X 8 cycles)
  Interventions: Drug: Adjuvant FOLFOX

INTERVENTIONS:
Drug: Adjuvant FL — 5-Fluorouracil 380 mg/m2, leucovorin 20 mg/m2 on D1-5 q 4 weeks X 4 cycles
  Other Names: fluorouracil, leucovorin
  Arms: Adjuvant FL
Drug: Adjuvant FOLFOX — oxaliplatin 85 mg/m2, leucovorin 200 mg/m2 on D1, 5-Fluorouracil bolus 400 mg/m2 on D1, 5-Fluorouracil continuous infusion 2400 mg/m2 for 46 hours q 2 weeks X 8 cycles
  Other Names: fluorouracil, oxaliplatin, leucovorin
  Arms: Adjuvant FOLFOX

SUMMARY:
The purpose of this study is to evaluate the disease-free survival in patients with locally advanced rectal cancer treated with preoperative chemoradiotherapy with fluoropyrimidines and surgery followed by adjuvant combination chemotherapy with oxaliplatin/5-FU/Leucovorin vs 5-FU/Leucovorin.

DETAILED DESCRIPTION:
Preoperative chemoradiotherapy with fluoropyrimidines followed by surgery is one of the standard treatments for patients with locally advanced rectal cancer; however, the role of adjuvant chemotherapy is still controversial. The aim of this study is to investigate the efficacy of adjuvant FOLFOX for rectal cancer who underwent fluoropyrimidine based chemoradiotherapy and complete total mesorectal excision.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the rectum
2. Patients who treated with preoperative chemoradiation with fluoropyrimidines followed by curative surgery without microscopic residual tumor.
3. AJCC/UICC pathologic stages of ypT3-4 or ypN+
4. Curative surgery not less than 3 and not more than 8 weeks prior to randomization
5. No prior chemotherapy, radiotherapy and immunotherapy except preoperative chemoradiation for rectal cancer
6. ECOG PS 0-1
7. Adequate organ function
8. Informed Consent

Exclusion Criteria:

1. Macroscopic or microscopic evidence of remaining tumor
2. Any histologic feature other than adenocarcinoma or arisen from chronic inflammatory bowel disease
3. More than 8 weeks after curative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2014-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, Professor, Principal Investigator — Asan Medical Center
Locations (6):
- South Korea (6):
  - National Cancer Center, Goyang
  - Seoul National Unversity Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yeonsei University Hosptial, Seoul

REFERENCES:
- [Derived] Hong YS, Kim SY, Lee JS, Nam BH, Kim KP, Kim JE, Park YS, Park JO, Baek JY, Kim TY, Lee KW, Ahn JB, Lim SB, Yu CS, Kim JC, Yun SH, Kim JH, Park JH, Park HC, Jung KH, Kim TW. Oxaliplatin-Based Adjuvant Chemotherapy for Rectal Cancer After Preoperative Chemoradiotherapy (ADORE): Long-Term Results of a Randomized Controlled Trial. J Clin Oncol. 2019 Nov 20;37(33):3111-3123. doi: 10.1200/JCO.19.00016. Epub 2019 Oct 8. PMID 31593484
- [Derived] Hong YS, Nam BH, Kim KP, Kim JE, Park SJ, Park YS, Park JO, Kim SY, Kim TY, Kim JH, Ahn JB, Lim SB, Yu CS, Kim JC, Yun SH, Kim JH, Park JH, Park HC, Jung KH, Kim TW. Oxaliplatin, fluorouracil, and leucovorin versus fluorouracil and leucovorin as adjuvant chemotherapy for locally advanced rectal cancer after preoperative chemoradiotherapy (ADORE): an open-label, multicentre, phase 2, randomised controlled trial. Lancet Oncol. 2014 Oct;15(11):1245-53. doi: 10.1016/S1470-2045(14)70377-8. Epub 2014 Sep 4. PMID 25201358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 screening failure due to raised carcinoembryonic antigen concentration
Groups:
- Adjuvant Fluorouracil +Leucovorin: FL (5-FU 380 mg/m2, leucovorin 20 mg/m2 on D1-5 q 4 weeks X 4 cycles)
  Adjuvant FL: 5-Fluorouracil 380 mg/m2, leucovorin 20 mg/m2 on D1-5 q 4 weeks X 4 cycles
Period: Overall Study
Arm/Group | Adjuvant Fluorouracil +Leucovorin | Adjuvant FOLFOX
Started | 161 | 160
Completed | 149 | 146
Not Completed | 12 | 14
Not completed — Withdrawal by Subject | 12 | 10
Not completed — Ineligible | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjuvant Fluorouracil +Leucovorin | Adjuvant FOLFOX | Total
Number analyzed (Participants) | 161 | 160 | 321
Age, Continuous [Median (Full Range); unit: years] | 54 [25 to 79] | 55 [27 to 81] | 54.5 [25 to 81]
Age, Customized [Count of Participants; unit: Participants]
  Aged 65 years or older | 24 | 31 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 42 | 87
  Male | 116 | 118 | 234
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Scale 0=Fully active, able to carry on all pre-disease performance without restriction;
  1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work;
  Participants
    0 | 30 | 26 | 56
    1 | 131 | 134 | 265
Distance of the primary tumour from the anal verge [Count of Participants; unit: Participants]
  ≤4 cm | 45 | 48 | 93
  >4 and ≤8 cm | 89 | 81 | 170
  >8 cm | 27 | 31 | 58
Tumor differentiation [Count of Participants; unit: Participants]
  Well differentiated | 20 | 13 | 33
  Moderately differentiated | 130 | 133 | 263
  Poorly differentiated/signet ring cell/mucinous | 9 | 11 | 20
  Undetermined | 2 | 3 | 5
Preoperative radiotherapy Dose [Median (Full Range); unit: cGY] | 5000 [5000 to 5040] | 5000 [5000 to 5040] | 5000 [5000 to 5040]
Preoperative radiotherapy duration [Median (Full Range); unit: weeks] | 5.0 [4.6 to 5.4] | 5.1 [4.9 to 5.7] | 5.05 [4.6 to 5.7]
Concurrent chemotherapy during preoperative radiotherapy [Count of Participants; unit: Participants]
  Fluorouracil with or without leucovorin | 108 | 107 | 215
  Capecitabine | 43 | 46 | 89
  Tegafur-uracil | 10 | 7 | 17
Concurrent chemotherapy during preoperative radiotherapy [Median (Full Range); unit: weeks] — Interval between end of preoperative chemoradiotherapy and surgery (weeks)
  weeks | 7.0 [6.0 to 8.0] | 7.0 [6.1 to 8.0] | 7.0 [6.0 to 8.0]
Type of surgery [Count of Participants; unit: Participants]
  Abdominoperineal resection | 24 | 24 | 48
  Low anterior resection | 135 | 135 | 270
  Hartmann's procedure | 2 | 1 | 3
Pathological T stage [Count of Participants; unit: Participants] — The post-neoadjuvant treatment tumor size which is determined by examining tissue removed during an operation.
  ypT0=No evidence of primary tumor; ypT1=Tumor invades the submucosa; ypT2=Tumor invades muscularis propria; ypT3=Tumor invades through the muscularis propria into pericolorectal tissues; ypT4=Tumor penetrates to the surface of the visceral peritoneum or directly invades or adheres to other organs or structures
  Participants
    ypT0 | 2 | 5 | 7
    ypT1 | 4 | 1 | 5
    ypT2 | 18 | 18 | 36
    ypT3 | 131 | 133 | 264
    ypT4 | 6 | 3 | 9
Pathological N stage [Count of Participants; unit: Participants] — The post-neoadjuvant treatment the extent of regional lymph node involvement which is determined by examining tissue removed during an operation.
  ypN0=No regional lymph node metastasis; ypN1a=Metastasis in one regional lymph node; ypN1b=Metastasis in 2-3 regional lymph nodes; ypN2a=Metastasis in 4-6 regional lymph nodes; ypN2b=Metastasis in seven or more regional lymph nodes
  Participants
    ypN0 | 65 | 58 | 123
    ypN1a | 30 | 42 | 72
    ypN1b | 38 | 25 | 63
    ypN2a | 19 | 29 | 48
    ypN2b | 9 | 6 | 15
yp stage [Count of Participants; unit: Participants] — stage grouping to assign an overall stage using ypT and N categories. Stage II(ypT3N0, ypT4N0), Stage III(ypTanyN1a, ypTany N1b, ypTanyN2a, ypTany N2b)
  Participants
    II | 65 | 58 | 123
    III | 96 | 102 | 198
Grade of tumour regression [Count of Participants; unit: Participants]
  Total regression | 2 | 5 | 7
  Near total regression | 22 | 31 | 53
  Moderate regression | 84 | 85 | 169
  Minimal or no regression | 52 | 38 | 90
  Unknown | 1 | 1 | 2
Lymphovascular invasion [Count of Participants; unit: Participants]
  Absent | 120 | 120 | 240
  Present | 41 | 37 | 78
  Unknown | 0 | 3 | 3
Time from surgery to randomisation (weeks) [Median (Full Range); unit: weeks] | 3.6 [3.1 to 4.6] | 3.4 [3.0 to 4.3] | 3.5 [3.0 to 4.6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Recurrence
Description: Disease-free survival will be measured as the time from the date of randomization to the date of disease relapse or death due to any cause. Using Cox-proportional hazard regression, the hazard ratio together with the 95% confidence interval will be reported, in addition to Kaplan-Meier estimates of the survival curves, including medians and rates with 95% confidence intervals. Intent-to-treat population included all randomised patients, and per-protocol population included patients who received at least 1 dose of chemotherapy without any violation of inclusion criteria
Time Frame: up to 3 years after completion of treatment
Population: intention-to-treat population (all randomised patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Fluorouracil +Leucovorin | Adjuvant FOLFOX
Number analyzed (Participants) | 161 | 160
Participants | 53 | 39
Statistical Analysis 1: Comparison: Adjuvant Fluorouracil +Leucovorin vs Adjuvant FOLFOX; Test type: Other; p = 0.047, t-test, 1 sided; Hazard Ratio (HR) = 0.657, 95% CI 2-sided [0.434 to 0.994]

2. Primary Outcome: Number of Participants With Disease Recurrence With Pathological Stage III
Description: as for outcome 1
Time Frame: up to 3 years after completion of treatment
Population: Among intention-to-treat population (all randomised patients), Patients with pathological stage III disease
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Fluorouracil +Leucovorin | Adjuvant FOLFOX
Number analyzed (Participants) | 96 | 102
Participants | 38 | 29
Statistical Analysis 1: Comparison: Adjuvant Fluorouracil +Leucovorin vs Adjuvant FOLFOX; Test type: Other; p = 0.040, t-test, 1 sided; Hazard Ratio (HR) = 0.602, 95% CI 2-sided [0.371 to 0.977]

3. Primary Outcome: Number of Participants With Disease Recurrence With Pathological Stage II
Description: as for outcome 1
Time Frame: up to 3 years after completion of treatment
Population: Among intention-to-treat population (all randomised patients), Patients with pathological stage II disease
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Fluorouracil +Leucovorin | Adjuvant FOLFOX
Number analyzed (Participants) | 65 | 58
Participants | 15 | 10
Statistical Analysis 1: Comparison: Adjuvant Fluorouracil +Leucovorin vs Adjuvant FOLFOX; Test type: Other; p = 0.47, t-test, 1 sided; Hazard Ratio (HR) = 0.744, 95% CI 2-sided [0.334 to 1.657]

4. Secondary Outcome: Death Rate
Description: overall survival was defined as the time from randomisation to death. We used the Kaplan-Meier method to estimate disease-free and overall survival. Patients were censored at the last follow-up if they were alive and free from disease recurrence. We used the log-rank test to compare the two survival distributions. We estimated crude and stratified hazard ratios (HRs) and their corresponding 95% CIs using the Cox proportionalhazards regression model.
Time Frame: Up to 3 years after completion of treatment.
Population: intention-to-treat population (all randomised patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Fluorouracil +Leucovorin | Adjuvant FOLFOX
Number analyzed (Participants) | 161 | 160
Participants | 21 | 10
Statistical Analysis 1: Comparison: Adjuvant Fluorouracil +Leucovorin vs Adjuvant FOLFOX; Test type: Other; p = 0.036, t-test, 1 sided; Hazard Ratio (HR) = 0.456, 95% CI 2-sided [0.215 to 0.970]

5. Secondary Outcome: Pattern of Recurrence
Description: After the completion of study treatment, chest radiography and measurement of carcinoembryonic antigen were done every 3 months for the fi rst 2 years and every 6 months thereafter. Abdominopelvic CT scans were done every 6 months and chest CT scans annually. Colonoscopy was scheduled at 1 year, 3 years, and 5 years from the date of surgery. Local recurrence was defined as any clinically proven tumour relapse within the pelvis or perineum. Distant metastasis was defined as relapse at any other site rather than local recurrence. We regarded any local or distant recurrence as a disease recurrence event. Disease recurrence was judged by the investigators with no central review.
Time Frame: the time from the date of randomization to the date of disease relapse, , assessed up to 5 years
Population: intention-to-treat population (all randomised patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Fluorouracil +Leucovorin | Adjuvant FOLFOX
Number analyzed (Participants) | 161 | 160
Participants
  Any event | 53 | 39
  Local recurrence | 12 | 5
  Distant metastasis | 44 | 35
  Lung | 29 | 24
  Liver | 15 | 8
  Lymph node | 10 | 6
  Bone | 4 | 2
  Peritoneum | 1 | 1
  Other* | 2 | 2

ADVERSE EVENTS:
Time Frame: 3 years
Description: 12 patients in the fluorouracil plus leucovorin group and 10 in the FOLFOX group were not received the planned treatment because of withdrawal. 4 patient in the FOLFOX group were not received the planned treatment because of ineligible.
  Death was assessed for all randomized participants. Adverse Events were assessed for all treated participants.
Groups:
- Fluorouracil+Leucovorin Group: FL (5-FU 380 mg/m2, leucovorin 20 mg/m2 on D1-5 q 4 weeks X 4 cycles) Adjuvant FL: 5-Fluorouracil 380 mg/m2, leucovorin 20 mg/m2 on D1-5 q 4 weeks X 4 cycles
- FOLFOX Group: FOLFOX (oxaliplatin 85 mg/m2, leucovorin 200 mg/m2 on D1, 5-FU bolus 400 mg/m2 on D1, 5-FU infusion 2400 mg/m2 for 46 hours q 2 weeks X 8 cycles) Adjuvant FOLFOX: oxaliplatin 85 mg/m2, leucovorin 200 mg/m2 on D1, 5-Fluorouracil bolus 400 mg/m2 on D1, 5-Fluorouracil continuous infusion 2400 mg/m2 for 46 hours q 2 weeks X 8 cycles
Arm/Group | Fluorouracil+Leucovorin Group | FOLFOX Group
All-Cause Mortality (participants affected / at risk) | 21/161 | 10/160
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/146
Other Adverse Events (participants affected / at risk) | 149/149 | 146/146
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluorouracil+Leucovorin Group (N=149) | FOLFOX Group (N=146)
Leucopenia (Blood and lymphatic system disorders) | 33 | 47
neutropenia (Blood and lymphatic system disorders) | 68 | 102
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 38
Anemia (Blood and lymphatic system disorders) | 3 | 3
Fatigue (General disorders) | 26 | 41
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 18
Nausea (Gastrointestinal disorders) | 56 | 78
Vomiting (Gastrointestinal disorders) | 17 | 19
Stomatitis (Gastrointestinal disorders) | 63 | 47
Diarrhea (Gastrointestinal disorders) | 38 | 49
Allergic reaction (Immune system disorders) | 1 | 3
Sensory neuropathy (Nervous system disorders) | 8 | 103

LIMITATIONS AND CAVEATS:
not specific

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No